CLINICAL TRIAL: NCT02598583
Title: An Open-Label, Intrapatient, Dose-Escalation Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of ALXN1210 Administered Intravenously to Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Dose-Escalation Study of ALXN1210 IV in Participants With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-103
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: PNH
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; complement inhibitor
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Participants were administered ALXN1210 900 mg.
  In the Extension period participants continued at the same dose and frequency as the Primary Evaluation Period.
  Interventions: Biological: ALXN1210
- Cohort 2 (Experimental): Participants were administered ALXN1210 1800 mg.
  In the Extension period participants continued at the same dose and frequency as the Primary Evaluation Period.
  Interventions: Biological: ALXN1210

INTERVENTIONS:
Biological: ALXN1210 — Participants were administered ravulizumab as an IV infusion every 4 weeks.

SUMMARY:
This study evaluated the safety, tolerability, efficacy, pharmacokinetics, pharmacodynamics, and immunogenicity of multiple intravenous (IV) doses of ALXN1210 administered to participants with PNH who have not previously been treated with complement inhibitor.

DETAILED DESCRIPTION:
The data presented is up to the Primary Completion date of the study and is for the 24-week Primary Evaluation period. The study also includes an Extension Period of up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. PNH diagnosis confirmed by documented high-sensitivity flow cytometry
3. Documented meningococcal vaccination not more than 3 years prior to dosing
4. Female participants of childbearing potential used highly effective contraception starting at screening and continuing until at least 24-weeks after the last dose of ALXN1210
5. Willing and able to give written informed consent and comply with the study visit schedule

Exclusion Criteria:

1. Treatment with a complement inhibitor at any time
2. Females who were pregnant, breastfeeding or who had a positive pregnancy test at screening or Day 1
3. Participation in an interventional clinical study within 30 days before initiation of dosing on Day 1, or use of any experimental therapy within 30 days prior to dosing on Day 1, or within 5 half-lives of the product, whichever is greater
4. History of allergy to excipients of ALXN1210 or known allergy to Chinese hamster ovary cell proteins
5. Inability to comply with study requirements
6. History of any clinically significant cardiac, hepatic, immunologic, pulmonary, or rheumatoid disease that, in the Investigator's judgment, would preclude participation
7. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, made the participant unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexion Pharmaceuticals, Inc., Study Director — Alexion Pharmaceuticals, Inc.
Locations (4):
- Australia (2):
  - Clinical Trial Site, Liverpool, New South Wales
  - Clinical Trial Site, Woolloongabba, Queensland
- South Korea (2):
  - Clinical Trial Site, Seoul
  - Clinical Trial Site, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Roth A, Rottinghaus ST, Hill A, Bachman ES, Kim JS, Schrezenmeier H, Terriou L, Urbano-Ispizua A, Wells RA, Jang JH, Kulasekararaj AG, Szer J, Aguzzi R, Damokosh AI, Shafner L, Lee JW. Ravulizumab (ALXN1210) in patients with paroxysmal nocturnal hemoglobinuria: results of 2 phase 1b/2 studies. Blood Adv. 2018 Sep 11;2(17):2176-2185. doi: 10.1182/bloodadvances.2018020644. PMID 30171081
- See also: Ravulizumab (ALXN1210) in patients with paroxysmal nocturnal hemoglobinuria: results of 2 phase 1b/2 studies — https://www.ncbi.nlm.nih.gov/pubmed/?term=Ravulizumab+(ALXN1210)+in+patients+with+paroxysmal+nocturnal+hemoglobinuria%3A+results+of+2+phase+1b%2F2+studies

RESULTS

PARTICIPANT FLOW:
Groups:
- ALXN1210 Cohort 1: Induction phase: a) 400 milligram (mg) on Day 1 and Day 8, 600 mg on Day 15; or b) 600 mg on Day 1, 600 mg on Day 15 Maintenance phase: the first of 5 doses of 900 mg on Day 29 and every 4 weeks thereafter
- ALXN1210 Cohort 2: Induction phase: 600 mg on Day 1, 900 mg on Day 15 Maintenance phase: the first of 5 doses of 1800 mg on Day 29 and every 4 weeks thereafter
Period: Primary Evaluation Period
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Started | 6 | 7
Completed (Completed 169-day Primary Evaluation Period.) | 6 | 7
Not Completed | 0 | 0
Period: Extension Period
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2 | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.87) | 43.6 (13.48) | 42.4 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 6 | 12
  White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change In Lactate Dehydrogenase (LDH) Levels From Baseline To Day 169
Description: Baseline was defined as the average of all available assessments prior to first ALXN1210 infusion.
Time Frame: Baseline, Day 169
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 LDH measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change | -85.952 (3.1897) | -84.736 (3.7736)

2. Secondary Outcome: Percent Change In Free Hemoglobin Levels From Baseline To Day 169 And Day 1821
Description: Baseline was defined as the last non-missing assessment value prior to the first ALXN1210 infusion.
Time Frame: Baseline, Day 169, Day 1821
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 free hemoglobin measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change
  Day 169 | -22.335 (42.2249) | -43.969 (24.7674)
  Day 1821: number analyzed (Participants) | 5 | 4
  Day 1821 | -35.062 (30.9356) | 24.435 (178.7882)

3. Secondary Outcome: Percent Change In Haptoglobin Levels From Baseline To Day 169 And Day 1821
Description: Baseline was defined as the last non-missing assessment value prior to the first ALXN1210 infusion.
Time Frame: Baseline, Day 169, Day 1821
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 haptoglobin measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change
  Day 169 | 40.0000 (55.13620) | 17.1429 (45.35574)
  Day 1821: number analyzed (Participants) | 5 | 4
  Day 1821 | 72.0000 (144.81022) | 62.5000 (125.00000)

4. Secondary Outcome: Percent Change In Reticulocyte/Erythrocyte Count From Baseline To Day 169 And Day 1821
Description: Baseline was defined as the last non-missing assessment value prior to the first ALXN1210 infusion.
Time Frame: Baseline, Day 169, Day 1821
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 reticulocyte/erythrocyte count measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change
  Day 169 | -21.203 (14.1461) | 28.784 (54.2636)
  Day 1821: number analyzed (Participants) | 5 | 4
  Day 1821 | -32.736 (18.8997) | 9.763 (22.5892)

5. Secondary Outcome: Percent Change In Paroxysmal Nocturnal Hemoglobinuria (PNH) Red Blood Cell (RBC) Clones From Baseline To Day 169 And Day 1933
Description: Baseline was defined as the last non-missing assessment value prior to the first ALXN1210 infusion.
Time Frame: Baseline, Day 169, Day 1933
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 PNH RBC clones measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change
  Day 169 | 7.873 (19.3064) | 25.840 (62.9677)
  Day 1933: number analyzed (Participants) | 3 | 2
  Day 1933 | 15.927 (34.8796) | 13.960 (78.9414)

6. Secondary Outcome: Percent Change In D-dimer Levels From Baseline To Day 169 And Day 1821
Description: Baseline was defined as the last non-missing assessment value prior to the first ALXN1210 infusion.
Time Frame: Baseline, Day 169, Day 1821
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 D-dimer measurement post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
percent change
  Day 169 | -27.42 (40.015) | -0.49 (73.116)
  Day 1821: number analyzed (Participants) | 5 | 4
  Day 1821 | -12.74 (54.821) | 25.15 (43.861)

7. Secondary Outcome: Change In Clinical Manifestations Of PNH From Baseline To Day 169 And Day 1821
Description: Clinical manifestations are defined as fatigue, abdominal pain, dyspnea, dysphagia, chest pain, and erectile dysfunction (ED) by cohort. Improvement is defined as present at baseline and absent at Day 169 endpoint. Worsening is defined as absent at Baseline and present at Day 169 endpoint.
Time Frame: Baseline, Day 169, Day 1821
Population: The full analysis set included all enrolled participants who received at least 1 dose of ALXN1210 and who had a Baseline measurement with at least 1 clinical manifestation of PNH assessed post-first ALXN1210 dose. Data were summarized only for participants with assessment at Baseline and the specified time point. ED affects only male participants.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
Participants
  Fatigue: Day 169: Improved from Baseline | 1 | 1
  Fatigue: Day 169: Worsened from Baseline | 0 | 0
  Fatigue: Day 169: No Change/Not Applicable | 5 | 6
  Fatigue: Day 1821: number analyzed (Participants) | 5 | 4
  Fatigue: Day 1821: Improved from Baseline | 2 | 1
  Fatigue: Day 1821: Worsened from Baseline | 0 | 0
  Fatigue: Day 1821: No Change/Not Applicable | 3 | 3
  Abdominal pain: Day 169: Improved from Baseline | 0 | 3
  Abdominal pain: Day 169: Worsened from Baseline | 0 | 0
  Abdominal pain: Day 169: No Change/Not Applicable | 6 | 4
  Abdominal pain: Day 1821: number analyzed (Participants) | 5 | 4
  Abdominal pain: Day 1821: Improved from Baseline | 0 | 2
  Abdominal pain: Day 1821: Worsened from Baseline | 0 | 0
  Abdominal pain: Day 1821: No Change/Not Applicable | 5 | 2
  Dyspnoea: Day 169: Improved from Baseline | 2 | 1
  Dyspnoea: Day 169: Worsened from Baseline | 0 | 0
  Dyspnoea: Day 169: No Change/Not Applicable | 4 | 6
  Dyspnoea: Day 1821: number analyzed (Participants) | 5 | 4
  Dyspnoea: Day 1821: Improved from Baseline | 2 | 1
  Dyspnoea: Day 1821: Worsened from Baseline | 0 | 0
  Dyspnoea: Day 1821: No Change/Not Applicable | 3 | 3
  Dysphagia: Day 169: Improved from Baseline | 0 | 1
  Dysphagia: Day 169: Worsened from Baseline | 0 | 0
  Dysphagia: Day 169: No Change/Not Applicable | 6 | 6
  Dysphagia: Day 1821: number analyzed (Participants) | 5 | 4
  Dysphagia: Day 1821: Improved from Baseline | 0 | 0
  Dysphagia: Day 1821: Worsened from Baseline | 0 | 0
  Dysphagia: Day 1821: No Change/Not Applicable | 5 | 4
  Chest pain: Day 169: Improved from Baseline | 0 | 2
  Chest pain: Day 169: Worsened from Baseline | 0 | 0
  Chest pain: Day 169: No Change/Not Applicable | 6 | 5
  Chest pain: Day 1821: number analyzed (Participants) | 5 | 4
  Chest pain: Day 1821: Improved from Baseline | 0 | 1
  Chest pain: Day 1821: Worsened from Baseline | 0 | 0
  Chest pain: Day 1821: No Change/Not Applicable | 5 | 3
  ED: Day 169: Improved from Baseline | 1 | 0
  ED: Day 169: Worsened from Baseline | 0 | 0
  ED: Day 169: No Change/Not Applicable | 5 | 7
  ED: Day 1821: number analyzed (Participants) | 4 | 1
  ED: Day 1821: Improved from Baseline | 1 | 0
  ED: Day 1821: Worsened from Baseline | 0 | 0
  ED: Day 1821: No Change/Not Applicable | 3 | 1

8. Secondary Outcome: Area Under The Serum Concentration-versus-time-curve From Time 0 (Dosing) To The Last Quantifiable Concentration (AUCt) At Day 1
Description: AUCt reported in hours*microgram/milliliter (h*ug/mL).
Time Frame: Day 1
Population: Pharmacokinetics (PK) Analysis Set: all participants who had sufficient serum concentration data to enable the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
h*ug/mL | 14273.95 (4907.438) | 42366.62 (3710.120)

9. Secondary Outcome: AUCt/ Dose-normalized (D) At Day 1
Time Frame: Day 1
Population: PK Analysis Set: all participants who had sufficient serum concentration data to enable the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: h*ug/mL/mg
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
h*ug/mL/mg | 35.68 (12.269) | 70.61 (6.184)

10. Secondary Outcome: Area Under The Serum Concentration-versus-time-curve From Time 0 (Dosing) To The End Of The Dosing Interval (AUCtau) At Day 141
Time Frame: Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
h*ug/mL | 216515.22 (68099.982) | 217936.47 (31023.979)

11. Secondary Outcome: AUCtau/D At Day 141
Time Frame: Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ug/mL/mg
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
h*ug/mL/mg | 240.57 (75.667) | 242.15 (34.471)

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) At Day 1 And Day 141
Time Frame: Day 1 and Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
ug/mL
  Day 1 | 114.00 (15.556) | 203.50 (10.279)
  Day 141 | 514.00 (147.078) | 512.25 (64.958)

13. Secondary Outcome: Cmax/D At Day 1 And Day 141
Time Frame: Day 1 and Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ug/mL/mg
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
ug/mL/mg
  Day 1 | 0.29 (0.039) | 0.34 (0.017)
  Day 141 | 0.57 (0.163) | 0.57 (0.072)

14. Secondary Outcome: Concentration At The End Of The Dosage Interval (Ctrough) At Day 1 And At Day 141
Time Frame: Day 1 and Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
ug/mL
  Day 1 | 73.25 (18.173) | 80.50 (6.541)
  Day 141 | 243.50 (126.572) | 204.00 (56.586)

15. Secondary Outcome: Time To Maximum Observed Serum Concentration (Tmax) At Day 1 And Day 141
Time Frame: Day 1 and Day 141
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 2 | 4
h
  Day 1 | 2.38 (2.404) | 1.88 (0.957)
  Day 141 | 4.03 (0.035) | 2.40 (1.124)

16. Secondary Outcome: Percent Change In Chicken Red Blood Cell (cRBC) Hemolysis From Baseline To Day 1709
Time Frame: Baseline, Day 1709
Population: Pharmacodynamics (PD) Analysis Set: all participants who had a measurement both before and after the first dose of ravulizumab.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 5 | 5
percent change | -72.316 (19.0919) | -97.314 (3.2298)

17. Secondary Outcome: Percent Change In Free Complement Component 5 (C5) Concentration From Baseline To Day 1709
Time Frame: Baseline, Day 1709
Population: PD Analysis Set: all participants who had a measurement both before and after the first dose of ravulizumab.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 5 | 5
percent change | -99.839 (0.0130) | -99.802 (0.0950)

18. Secondary Outcome: Percent Change In Total C5 Concentration From Baseline To Day 1709
Time Frame: Baseline, Day 1709
Population: PD Analysis Set: all participants who had a measurement both before and after the first dose of ravulizumab.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 5 | 5
percent change | 65.852 (31.2054) | 86.676 (24.6721)

19. Secondary Outcome: Participants Experiencing Antidrug Antibodies (ADAs)
Time Frame: Day 1821
Population: Immunogenicity Analysis Set: all participants who had an ADA sample both before and after the first dose of ravulizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

20. Post Hoc Outcome: Percent Change In LDH Levels From Baseline To Day 1821
Description: Baseline was defined as the average of all available assessments prior to first ALXN1210 infusion.
Time Frame: Baseline, Day 1821
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
Number analyzed (Participants) | 5 | 4
percent change | -86.244 (4.7348) | -84.413 (3.6473)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 1957
Arm/Group | ALXN1210 Cohort 1 | ALXN1210 Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1210 Cohort 1 (N=6) | ALXN1210 Cohort 2 (N=7)
Meningococcal infection (Infections and infestations) | 0 | 1
Parvovirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1210 Cohort 1 (N=6) | ALXN1210 Cohort 2 (N=7)
Headache (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Hordeolum (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2
Laryngitis (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Parvovirus infection (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Chlamydial infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Laryngopharyngitis (Infections and infestations) | 0 | 1
Nipple infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oophoritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Face oedema (General disorders) | 0 | 1
Puncture site pain (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes